CLINICAL TRIAL: NCT04031352
Title: Investigation of Factors Affecting Children's Attitudes Towards Peers With Disability
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, ALI KITIS, PROFESSOR, Pamukkale University
Other Study IDs: 17531
Record Dates: First submitted 2019-07-15; First posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Disability Physical
Keywords: attitude; CATCH; children; disability; peers
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: implementation of CATCH scale — subject completed the CATCH scale

SUMMARY:
Children with disabilities can be exposed to stigma and discrimination because of poor attitudes. The role of peer is crucial for development of disabled children.

The aim of the study was to investigate the attitudes of children towards their peers with disabilities and to identify factors associated with them.

1305 elementary school students included to the study. The students participating in the study, 48.9% (534) were female, 51.1% (558) were male. The Chedoke-McMaster Attitudes towards Children with Handicaps (CATCH) scale was used to investigate the children's attitudes.

DETAILED DESCRIPTION:
* Being important in terms of epidemiological investigation.
* Giving new results from society with different cultural and national characteristics.
* Investigating the three components of the CATCH.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were being a student of elementary school, being aged between 11-15 years and being volunteer.

Exclusion Criteria:

* Students who had a congenital or acquired disability or a handicap and who did not complete the scale were excluded.

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 1305 elementary school students (aged 11-14 years and grades 5-8) included to the study from 6 public and 2 private schools. The students participating in the study, 48.9% (534) were female, 51.1% (558) were male.
Sampling Method: Non-Probability Sample
Enrollment: 1305 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2018-02-18 (Actual); Study Completion 2018-06-16 (Actual)

PRIMARY OUTCOMES:
CATCH | one year
  The Chedoke-McMaster Attitudes towards Children with Handicaps Scale The CATCH scale contains 36 items. It is divided into three components. First, the affective component contains 12 items that focus on feelings towards people with disabilities. Second, the cognitive component contains 12 items that focus on beliefs towards people with disabilities. Third, the behavioural component contains 12 items that focus on behaviours towards people with disabilities. The CATCH scale was designed for children aged 9-13 years. The highest possible mean score on the overall scale or in any component is 40. A high score represents a more positive attitude

CONTACTS AND LOCATIONS:
Overall Officials: ALI KITIS, PROF, Study Chair — Pamukkale University; OZGE MINE YILMAZ, MSC, Principal Investigator — Pamukkale University; HANDE USTA, PHDc, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided